CLINICAL TRIAL: NCT04552782
Title: PTSD, AUD, and Interpersonal Conflict: Within-person Associations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Dakota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Sioux Falls VA Health Care System (U.S. Federal Agency); Bay Pines VA Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R01MH122954 (NIH)
Record Dates: First submitted 2020-09-10; First posted 2020-09-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Stress Disorders, Post-Traumatic; Alcoholism
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcohol Cognitive Bias Modification (CBM) + PTSD CBM (Experimental)
  Interventions: Behavioral: Alcohol CBM; Behavioral: PTSD CBM
- Alcohol CBM + PTSD Sham (Experimental)
  Interventions: Behavioral: Alcohol CBM; Behavioral: PTSD Sham
- Alcohol Sham + PTSD CBM (Experimental)
  Interventions: Behavioral: PTSD CBM; Behavioral: Alcohol Sham
- Alcohol Sham + PTSD Sham (Sham Comparator)
  Interventions: Behavioral: Alcohol Sham; Behavioral: PTSD Sham

INTERVENTIONS:
Behavioral: Alcohol CBM — Trains approach or avoidance responses to alcohol cues.
  Arms: Alcohol CBM + PTSD Sham; Alcohol Cognitive Bias Modification (CBM) + PTSD CBM
Behavioral: PTSD CBM — Trains approach or avoidance responses to trauma cues.
  Arms: Alcohol Cognitive Bias Modification (CBM) + PTSD CBM; Alcohol Sham + PTSD CBM
Behavioral: Alcohol Sham — Will not train approach or avoidance responses.
  Arms: Alcohol Sham + PTSD CBM; Alcohol Sham + PTSD Sham
Behavioral: PTSD Sham — Will not train approach or avoidance responses.
  Arms: Alcohol CBM + PTSD Sham; Alcohol Sham + PTSD Sham

SUMMARY:
The present study seeks to increase understanding of Alcohol Use Disorder (AUD) and Posttraumatic Stress Disorder (PTSD) among veterans, an important public health concern. We will study the effects of regulatory deficits and sleep disturbance on the dynamic course of PTSD and AUD. The study will investigate whether a short, computerized training in the laboratory will alter maladaptive response biases and reduce associations between sleep disturbance, affect and behavioral dysregulation, AUD symptoms, and PTSD symptoms in the real world.

ELIGIBILITY:
Inclusion Criteria:

* OIF/OEF/OND veterans
* At risk for PTSD (i.e., PCL-5 ≥33) and/or AUD (i.e., AUDIT ≥ 7 (women) ≥ 8 (men))

Exclusion Criteria:

* Psychosis or severe Alcohol Use Disorder that contraindicates participation (based on interview)
* Active suicidal or homicidal ideation that contraindicates participation (based on interview)
* [exclusion criteria removed 6/2022] - Severe risk for sleep apnea (a positive score in three categories of the Berlin Questionnaire), or reported treatment for sleep apnea

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Alcohol Use Disorder Symptoms | 2 years
  These are experience sampling items derived from Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
Rate of PTSD Symptoms | 2 years
  These are experience sampling items derived from the PTSD Checklist from DSM-5 (PCL-5).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bay Pines VA Health Care System, Bay Pines, Florida
  - Sioux Falls VA Health Care System, Sioux Falls, South Dakota
  - The University of South Dakota, Vermillion, South Dakota